CLINICAL TRIAL: NCT00585429
Title: Kidney Disease in Advanced Liver Disease Patients: A Study of Kidney Damage by a Urinary Cytokine/Chemokine Multiplex Assay
Brief Title: Evaluation of Kidney Disease in Liver Transplant Recipients
Status: Withdrawn | Type: Observational
Why Stopped: key personnel left institution
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: H-2006-0335
Record Dates: First submitted 2007-12-26; First posted 2008-01-03 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Kidney Disease; Liver Transplantation
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: ESLD subjects on active liver transplant waiting list
- 2: Subjects post-liver transplant with good liver function
- 3: Subjects without liver disease undergoing kidney biopsy for diagnostic purposes

SUMMARY:
A non-invasive urinary test that detects kidney injuries in liver transplant (LT) candidates would be useful for monitoring of kidney damage. Particularly, the ability to predict irreversibility of such renal damage or progressive nature of renal disease in LT candidates would be of importance to determine the need for dual kidney-liver transplantation (KLT) versus LT alone. We will correlate kidney histology with cytokine/chemokine profile expression in the urine as a potentially useful noninvasive diagnostic tool.

ELIGIBILITY:
Inclusion Criteria:

* Subjects on the liver transplant wait list, subjects who have received a liver transplant at least 6 months prior to enrollment, or subjects who have normal liver function and are about to undergo kidney biospy for diagnostic purposes.

Exclusion Criteria:

* Contraindication to kidney biopsy
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects on the liver transplant wait list, subjects who have received a liver transplant at least 6 months prior to enrollment, or subjects who have normal liver function and are about to undergo kidney biospy for diagnostic purposes.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2006-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To determine the value of urinary levels of chemokines in the distinction between types of kidney disease in the setting of liver failure | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States